CLINICAL TRIAL: NCT02563483
Title: A Yoga and Compassion Meditation Program Improve Quality of Life and Self-compassion in Family Caregivers of Alzheimer's Disease Patients: a Randomized Controlled Trial
Brief Title: Yoga for Family Caregivers of Alzheimers Disease Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, JGalduroz, MD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: yoga caregivers
Record Dates: First submitted 2015-09-28; First posted 2015-09-30 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Stress; Anxiety; Compassion
Keywords: caregivers; anxiety; depression; yoga; meditation; stress
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga and compassion meditation program (Experimental): The duration of this group was 8 weeks. The program included sessions 3 times per week, with each session lasting 1 hour and 15 minutes. The volunteers performed yoga classes composed of "asana" (poses), "pranayama" (breathing exercise) and meditation.
  Interventions: Behavioral: yoga and compassion meditation program
- control (No Intervention): this group was a non treatment group.

INTERVENTIONS:
Behavioral: yoga and compassion meditation program — 25 min of physical exercise, holding each pose (stretching exercise) for an average of 1 min and 30 s; 25 min of breathing exercises and 25 min of meditation.
  Arms: Yoga and compassion meditation program

SUMMARY:
This study evaluates the effects of the practice of yoga in combination with compassion meditation on the quality of life, attention, vitality and self-compassion of family caregivers of patients with Alzheimer's disease.

DETAILED DESCRIPTION:
Alzheimer's disease is a progressive brain disorder that involves the loss of reasoning, memory, language and the ability to live independently. Thus, patients who suffer from this disease often require care from another person and must adapt to ensure their health, functional capacity and safety. Caregivers have a poor quality of life due to the physical and psychological burden of caregiving. Such physical, psychological, social and financial burden can increase the risk of death. Within this scenario, techniques such as yoga and meditation have emerged as low-cost interventions that offer little or no risk to the practitioners. Yoga seeks to develop health and attention through physical postures, breathing exercises and formal meditative practices.

ELIGIBILITY:
Inclusion Criteria:

* be a family caregiver of Alzheimer disease patient
* age over 18 years
* completed at least the primary education level
* at least at the phase of stress resistance according to Lipp's Inventory of Stress Symptoms for adults

Exclusion Criteria:

* patient with asthma or chronic obstructive pulmonary disease (COPD)
* alcohol use (more than 5 drinks per week) or use of drugs-of-abuse;
* suffer from Cushing's syndrome
* under treatment with topical, nasal or any form of steroids within the last 30 days
* practice yoga, meditation or similar techniques

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-09; Primary Completion 2008-02 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
change in cortisol | baseline, 8 weeks
  Saliva samples were collected for analysis of cortisol

SECONDARY OUTCOMES:
change in stress | baseline, 8 weeks
  Lipp Stress Inventory
change in depression | baseline, 8 weeks
  Beck Depression Inventory
change in anxiety | baseline, 8 weeks
  Beck Anxiety Inventory
change in quality of life | baseline, 8 weeks
  WHOQOL-bref (World Health Organization Quality of Life Questionnaire with 26 questions)
change in vitality | baseline, 8 weeks
  Subjective Vitality Scales
change in attention | baseline, 8 weeks
  Mindfulness Attention Awareness Scale
change in self-compassion | baseline, 8 weeks
  Self-Compassion Scale

REFERENCES:
- [Background] Danucalov MA, Kozasa EH, Ribas KT, Galduroz JC, Garcia MC, Verreschi IT, Oliveira KC, Romani de Oliveira L, Leite JR. A yoga and compassion meditation program reduces stress in familial caregivers of Alzheimer's disease patients. Evid Based Complement Alternat Med. 2013;2013:513149. doi: 10.1155/2013/513149. Epub 2013 Apr 18. PMID 23690846
- See also: A yoga and compassion meditation program reduces stress in familial caregivers of Alzheimer's disease patients — http://www.ncbi.nlm.nih.gov/pubmed/23690846